CLINICAL TRIAL: NCT03052296
Title: BIOTRONIK - A Prospective, National, Multi-centre, Post-market Registry to Assess the Clinical Performance of the Passeo-18 Lux Paclitaxel Releasing Balloon Catheter in Long Femoropopliteal Artery Lesions - III SPAIN
Brief Title: BIOLUX P-III SPAIN All-Comers Registry
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1603
Record Dates: First submitted 2017-02-02; First posted 2017-02-14 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Passeo-18 Lux DCB — The endovascular procedure is conducted as per the local standard practice and device instruction for use

SUMMARY:
The purpose of the BIOLUX P-III Spain registry is to further investigate the safety and clinical performance of the Passeo-18 Lux Drug Coated Balloon in the treatment of long atherosclerotic femoropoliteal artery lesions in daily clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* Subject must be willing to sign a Patient Data Release Form (PDRF) or Patient Informed Consent (PIC) where applicable
* Subject classified as Rutherford class 4, 5 or 6
* TASC C or D lesion(s) in the femoropopliteal artery
* Lesion length > 15 cm suitable for endovascular treatment treated with or scheduled to be treated with the Passeo-18 Lux drug releasing balloon

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Subject is currently participating in another investigational drug or device study that has not reached its primary endpoint yet.
* Subject is pregnant or planning to become pregnant during the course of the study.
* Rutherford class <4
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations).
* Intraprocedural decision not to proceed with the Passeo18 Lux DCB for any reason not related to the device (for instance blood flow limiting dissection after predilatation).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The BIOLUX P-III SPAIN registry will include subjects from an all-comers patient population with all subjects requiring revascularization of long femoropopliteal artery lesions with the Passeo-18 Lux DCB
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events (MAE) | 6 months
  A composite of freedom from device- and procedure-related mortality through 30 days, and freedom from major target limb amputation and clinically driven target lesion revascularization (TLR)
Freedom from clinically driven Target Lesion Revascularization (TLR) | 12 months
  Any re-intervention performed for ≥ 50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent clinical symptoms of the patient.)

SECONDARY OUTCOMES:
Freedom from clinically-driven target lesion revascularization (TLR) | 6 months
Freedom from clinically-driven target vessel revascularization (TVR) | 6 and 12 months
Primary Patency | 12 months
  defined as freedom from >50% restenosis in the target lesion as indicated by a duplex ultrasound peak systolic velocity ratio (PSVR) >2.5 or by visual assessment of an angiogram with no clinically driven re-intervention.
Freedom from MAE | 12 months
  Composite of freedom from device- and procedure-related mortality through 30 days, and freedom from major target limb amputation and clinically driven TLR
Change in mean Ankle Brachial Index (ABI) | 6 and 12 months
  Thigh or toe brachial index (TBI) may be used / performed if ABI is inadequate
Improvement in Rutherford classification compared to the pre-procedure Rutherford classification | 6 and 12 months
Amputation-free survival (AFS) including major, minor and overall AFS | 6 and 12 months
Pain score compared to the pre-procedure score | 6 and 12 months
Walking Impairment Questionnaire compared to the pre-procedure score | 6 and 12 months
Device success | Immediately upon procedure
  Successful delivery, inflation, deflation, and retrieval of the Passeo-18 Lux DCB.
Technical success | Immediately upon procedure
  Successful completion of the endovascular procedure and immediate morphological success with ≤ 50% residual diameter reduction of the treated lesion as determined by visual estimation.
Procedural success | Immediately upon discharge
  Procedural success is technical and device success without the occurrence of any MAE (as defined in the protocol) during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel de Gregorio, Principal Investigator — Hospital Clínico and University of Zaragoza
Locations (5):
- Spain (5):
  - Hospital Mataró, Barcelona
  - Hospital San Cecilio, Granada
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen de la Macarena, Seville
  - Hospital Clínico Lozano Blesa Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No